CLINICAL TRIAL: NCT06070792
Title: The Effect of Neuro Linguistic Program and Progressive Muscle Relaxation Exercises on Breastfeeding Success and Breastfeeding Self-efficacy After Caesarean Section
Brief Title: Neurolinguistic Programming, Progressive Muscle Relaxation Exercises, and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, Gaziantep University Health Sciences Enstıtute, Department of Nursing, Department of Obstetrics and Gynaecology Nursing, PhD., University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NLP, PMRE, AND BREASTFEEDING
Record Dates: First submitted 2023-09-19; First posted 2023-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NEUROLINGUISTIC PROGRAMMING; PROGRESSIVE MUSCLE RELAXATION EXERCISES; CAESAREAN SECTION
Keywords: NEURO LINGUISTIC PROGRAM; PROGRESSIVE MUSCLE RELAXATION EXERCISES; CAESAREAN SECTION; BREASTFEEDING SUCCESS; BREASTFEEDING SELF-EFFICACY

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NEURO LINGUISTIC PROGRAM (Experimental): first experimental group. It will be administered to primiparous mothers after caesarean section in the first 48 hours after the sixth postoperative hour, once every eight hours, for a total of six times. Each session will last 20 minutes.
  In the NLP application; firstly, the most frequently used visual, auditory and/or tactile representation system of the woman will be determined. Then, the internal and external reactions caused by the symptoms after caesarean section, her feelings and thoughts about her baby and breastfeeding will be combined with the anchoring technique. Then, with the swish technique, the existing negative emotions will be reduced and tried to be deleted from the most frequently used representation system. The woman's negative thoughts about breastfeeding will be changed in a positive direction with the belief change model.
  Interventions: Other: NEURO LINGUISTIC PROGRAM
- PROGRESSIVE MUSCLE RELAXATION EXERCISES (Experimental): second experimental group. It will be administered to primiparous mothers after caesarean section in the first 48 hours after the sixth postoperative hour, once every eight hours, for a total of six times. Each session will last 20 minutes.
  PMRE; All muscles of the body will be tried to be relaxed respectively with the commands given gradually.
  Interventions: Other: PROGRESSIVE MUSCLE RELAXATION EXERCISES
- control (No Intervention): The control group will not receive NLP or PMRE.

INTERVENTIONS:
Other: NEURO LINGUISTIC PROGRAM — NEURO LINGUISTIC PROGRAM
  Arms: NEURO LINGUISTIC PROGRAM
Other: PROGRESSIVE MUSCLE RELAXATION EXERCISES — PROGRESSIVE MUSCLE RELAXATION EXERCISES
  Arms: PROGRESSIVE MUSCLE RELAXATION EXERCISES

SUMMARY:
The effect of neuro linguistic program and progressive muscle relaxation exercises on breastfeeding success and breastfeeding self-efficacy after caesarean section.

DETAILED DESCRIPTION:
In this research, it is aimed to detemine the effect of neuro linguistic program and progressive muscle relaxation exercises on breastfeeding success and breastfeeding self-efficacy after caesarean section.

Sample size:

* There will be three groups in the study (two experimental groups and one control group).
* The sample size of the study is 99 people. The sample size will be divided into three and 33 people will be randomly assigned to each group.
* Experiment 1 group: neuro linguistic programme (NLP) group.
* Experiment 2 group: progressive muscle relaxation exercises (PMRE) group.
* Control group: non-intervention group

Data Collection Tools;

* Introductory Information Form,
* Breastfeeding Self-Efficacy Scale,
* Breastfeeding Charting System (LATCH)

Application time:

* NLP and PMRE interventions will be started at the sixth postoperative hour after caesarean section.
* Mothers who give birth by caesarean section are followed up in hospital for 48 hours and mothers are then discharged when their health condition improves. Therefore, data will be collected within 48 hours after caesarean section.
* NLP and PMRE groups will be started at the sixth postoperative hour, 3 times in 24 hours on the first day, 3 times in 24 hours on the second day, six times in total.
* Only NLP and PMRE will not be applied to the control group.
* Care and follow-up will be performed in parallel with the individuals in the experimental group.

Measurement time:

* Mothers will fill in the Introductory Information Form, Breastfeeding Self-Efficacy Scale, Breastfeeding Diagnosis and Assessment Measurement Tool (LATCH) before the application at the sixth postoperative hour.
* Then, in the first 24 hours, the necessary application will be performed once every eight hours according to the groups (for example, NLP application for experiment 1).
* At the end of 24th hour, Breastfeeding Self-Efficacy Scale and Breastfeeding Diagnosis and Assessment Measurement Tool (LATCH) will be completed.
* Then, in the second 24 hours, the interventions will be repeated once every eight hours.
* The total number of application sessions is six.
* NLP application will last 20 minutes each session and PMRE application will last 20 minutes each session.

ELIGIBILITY:
Inclusion Criteria:

* women who gave birth by caesarean section,
* primiparous,
* who are 19 years of age or older and 35 years of age or younger,
* who were born at 37 or more weeks of gestation,
* who had a singleton birth,
* whose caesarean section operation was performed with spinal anaesthesia,
* who do not have chronic diseases and any breast-related health problems .

Exclusion Criteria:

* mothers who did not meet the inclusion criteria,
* who wanted to leave the study voluntarily at any stage after being included in the study,
* who developed any health problems in themselves or their infants were excluded.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primiparous mothers giving birth by caesarean section for the first time
Enrollment: 99 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
BREASTFEEDING SUCCESS | immediately before the first application
  Breastfeeding Charting System (LATCH); The measurement tool has no cut-off point, and as the LATCH score increases, it is understood that the process is high. The maximum score that can be obtained is 10. The sum of lower scores indicates that the mother is dependent on help.
BREASTFEEDING SUCCESS | immediately after the third application (at the 24th hour after the first application)
  Breastfeeding Charting System (LATCH)
BREASTFEEDING SUCCESS | immediately after the sixth application (at the 48th hour after the first application)
  Breastfeeding Charting System (LATCH)
BREASTFEEDING SELF-EFFICACY | immediately before the first application
  Breastfeeding Self-Efficacy Scale; A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All are positive elements. The higher the score from the scale, the higher breastfeeding self-efficacy will be achieved.
BREASTFEEDING SELF-EFFICACY | immediately after the third application (at the 24th hour after the first application)
  Breastfeeding Self-Efficacy Scale
BREASTFEEDING SELF-EFFICACY | immediately after the sixth application (at the 48th hour after the first application)
  Breastfeeding Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilicli A, Gul S. The effect of neurolinguistic programming and progressive muscle relaxation exercises on breastfeeding success and breastfeeding self-efficacy: A randomized controlled trial. Explore (NY). 2024 Sep-Oct;20(5):103027. doi: 10.1016/j.explore.2024.103027. Epub 2024 Jul 2. PMID 39003935